CLINICAL TRIAL: NCT01079273
Title: An Open-Label Exploratory Clinical Study to Evaluate the Antibody and Cell Mediated Immunity of One Intramuscular Dose of MF59-Adjuvanted Egg-Derived, Inactivated Novel Swine Origin A/H1N1 Monovalent Subunit Influenza Virus Vaccine in Healthy Subjects Aged 18 to 60 Years
Brief Title: Clinical Study to Evaluate Antibody and Cell Mediated Immunity of A/H1N1 Influenza Vaccine in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: V111_06TP_OPERA; 2009-017141-58 (EudraCT Number)
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Influenza
Keywords: Influenza; Vaccines; A/H1N1; Influenza Vaccines
MeSH Terms: conditions — Influenza, Human | interventions — focetria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine (Active Comparator): All Subjects enrolled in this study will receive the study vaccine (single-arm)
  Interventions: Biological: egg-derived A/H1N1 pandemic influenza vaccine

INTERVENTIONS:
Biological: egg-derived A/H1N1 pandemic influenza vaccine — One 0.50 mL IM dose injection (7.5 µg of vaccine + 9.75 mg MF59)
  Other Names: Focetria™

SUMMARY:
The purpose of this study is explore the antibody and cell mediated immune responses to one injection of Focetria™ pandemic influenza vaccine in healthy adults aged 18-60 years.

DETAILED DESCRIPTION:
This will be a Phase IV open-label clinical profiling study. The population to be enrolled will consist of healthy adults aged 18-60 years. A total of approximately 60 subjects are planned for enrolment into this study.

Subjects enrolled in this study will receive 7.5 µg of vaccine + MF59 (9.75 mg/dose). Each subject will receive one 0.5 mL IM dose (deltoid muscle, non-dominant arm) of H1N1sw vaccine at Visit 1, after the blood draw. Up to 70 mL of blood will be drawn for CMI and antibody assessment from all subjects at all study visits.

Subjects will be requested to declare occurrence of influenza-related symptoms during the study period. Whenever appropriate, subjects might be asked to provide throat swab for viral typing. Subjects with laboratory confirmed H1N1sw influenza might be asked to provide one blood sample (70 mL) within 4 weeks after influenza resolution.

Although this study is not designed nor powered to draw conclusions regarding safety and tolerability, all subjects will be followed, but not analyzed, for safety throughout the study. After vaccination, all subjects will remain under medical supervision at the study site for 30 minutes to be monitored and evaluated for possible immediate hypersensitivity reactions. All study subjects will be instructed on the completion of diary cards to record local and systemic reactions for seven days, starting on the day of vaccination and continuing during the 6 following days. The same diary cards will additionally be used to collect any vaccine-related reactions and any changes in the subject's health (including any serious medical problems such as hospitalizations or any life-threatening medical problems) and any medications taken by the subject throughout the study. All serious adverse events and all adverse events will be recorded throughout the entire trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained;
* Males and females from 18 years to 60 years of age on the day of enrolment;
* Subjects in good health as determined by the outcome of medical history, physical assessment and clinical judgment by the Investigator;
* Subjects are able to comply with all study procedures and are available for all clinic visits scheduled in the study;
* Willingness to allow for blood samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

* Subjects who are not able to comprehend and to follow all required study procedures for the whole period of the study;
* Subjects with history or any illness that, in the opinion of the Investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study;
* Subjects with any serious chronic or progressive disease according to judgment of the Investigator (including, but not limited to malignant neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease);
* History of any anaphylaxis, serious vaccine reactions, or hypersensitivity to influenza viral proteins, to any excipients, and to eggs (including ovalbumin), and chicken proteins;
* Subjects who have had seasonal influenza vaccine or documented confirmed seasonal influenza disease within 2 weeks prior to Day 1;
* Receipt of another investigational agent within 4 weeks prior to enrolment, or before completion of the safety follow-up period in this or in another study; subjects unwilling to refuse participation in another clinical study throughout the end of this study;
* Subjects who received any other vaccines within 4 weeks prior to enrolment in this study or who are planning to receive any vaccine within 4 weeks from the study vaccines; the only exception being plain seasonal influenza vaccines which are allowed until 2 weeks before and over 2 weeks after the study vaccination;
* Subjects who have received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks or plan to receive these products during the full length of the study;
* Subjects with axillary temperature ≥ 38°C (≥ 100.4°F) or oral temperature ≥ 38.5°C (≥ 101.3°F) within 3 days of intended study vaccination;
* Known or suspected impairment/alteration of immune function, for example resulting from:

  1. receipt of immunosuppressive therapy such as systemic corticosteroids known to be associated with the suppression of hypothalamic-pituitary-adrenal (HPA) axis (10 mg/day of prednisone or its equivalent) or chronic use of inhaled high-potency corticosteroids (e.g. budesonide 800µg/day or fluticasone 750µg/day) within 60 days prior to Visit 1,
  2. cancer chemotherapy within 5 years,
  3. receipt of immunostimulants within 60 days prior to Visit 1,
  4. history of HIV infection or HIV-related disease;
* History of progressive or severe neurological disorders (including Guillain-Barré syndrome and convulsions, but excluding febrile convulsions);
* History of or clinically suspected developmental delay;
* Bleeding diathesis;
* Surgery planned during the study period that in the Investigator's opinion would interfere with the study;
* Female subjects who are pregnant or nursing (breastfeeding) mothers, or females of childbearing potential who are sexually active and have not used any of the "acceptable contraceptive methods" for the 2 months before entering the study or do not plan to use them up to the end of the study;
* Members of the research staff who have direct access to any study documents containing subject information.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2009-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Antibody and cell mediated immune responses to one 0.50 mL IM injection of egg-derived Focetria™ pandemic influenza vaccine in terms of quality and quantity of the antigen-specific T- and B-cell response | On day 8, 22, 202 after vaccination
  Cell Mediated Immunity (CMI) assessed by frequencies and fold increases of antigen-specific CD4+ T-cells and B-lymphocytes on Day 0,8,22,202.
  Immunogenicity, i.e. Haemagglutination Inhibition (HI), Single Radial Haemolysis (SRH) and Microneutralization (MN), assessed as follows:
  1. Geometric mean titer (GMT)/Geometric mean area (GMA) on Day 0,8,22,202.
  2. Geometric mean ratio (GMR) at each time-point vs. Day 0.
  3. Percentage of subjects achieving seroconversion or significant increase on Day 8,22,202.
  4. Percentage of subjects with HI (or MN) titer≥40 and SRH≥25 mm2 on Day 0,8,22,202.

SECONDARY OUTCOMES:
Antibody responses to one injection of egg-derived Focetria™ pandemic influenza vaccine according to CHMP criteria | On day 8, 22, 202 after vaccination
  In the interpretation of HI immunogenicity results, the following Committee for Medicinal Products for Human Use (CHMP) criteria (CPMP/BWP/214/96) for healthy adults will be taken in consideration:
  * The proportion of subjects achieving seroconversion or significant increase in HI antibody titer should be > 40%
  * Mean geometric increase should be > 2.5
  * The proportion of subjects achieving an HI titer ≥ 40 should be > 70%.
Safety and tolerability | Within 30 minutes after vaccination (Day 0) and on day 8, 22 and 202 after vaccination
  A medical history will be obtained and physical assessment performed for each subject entered into the study at the time of enrolment and then, a brief physical assessment after every subsequent visit. All subjects will be followed for safety throughout the study. All serious adverse events and all adverse events will be collected throughout the entire trial using diary cards.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Laghi Pasini, MD, Principal Investigator — Azienda Ospedaliera Universitaria Senese; Laura Michellini, Study Chair — Opera CRO, a TIGERMED Group Company; Fabio Montanaro, DSc, Study Director — Opera CRO, a TIGERMED Group Company
Locations (1):
- Azienda Ospedaliera Universtaria Senese, Siena, Italy

REFERENCES:
- [Result] Faenzi E, Zedda L, Bardelli M, Spensieri F, Borgogni E, Volpini G, Buricchi F, Pasini FL, Capecchi PL, Montanaro F, Belli R, Lattanzi M, Piccirella S, Montomoli E, Ahmed SS, Rappuoli R, Del Giudice G, Finco O, Castellino F, Galli G. One dose of an MF59-adjuvanted pandemic A/H1N1 vaccine recruits pre-existing immune memory and induces the rapid rise of neutralizing antibodies. Vaccine. 2012 Jun 8;30(27):4086-94. doi: 10.1016/j.vaccine.2012.04.020. Epub 2012 Apr 19. PMID 22521851
- [Derived] Ahmed SS, Volkmuth W, Duca J, Corti L, Pallaoro M, Pezzicoli A, Karle A, Rigat F, Rappuoli R, Narasimhan V, Julkunen I, Vuorela A, Vaarala O, Nohynek H, Pasini FL, Montomoli E, Trombetta C, Adams CM, Rothbard J, Steinman L. Antibodies to influenza nucleoprotein cross-react with human hypocretin receptor 2. Sci Transl Med. 2015 Jul 1;7(294):294ra105. doi: 10.1126/scitranslmed.aab2354. PMID 26136476